CLINICAL TRIAL: NCT02214251
Title: The Electrophysiological Investigation of Higher Level Neural Manifestations of Freezing of Gait in Parkinson's Disease Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, Chon-Haw Tsai, The chief, Department of Neurology, China Medical University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CMUH103-REC2-017
Record Dates: First submitted 2014-08-08; First posted 2014-08-12 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Parkinson's Disease; Freezing of Gait
Keywords: Parkinson's disease; freezing of gait; movement disorders; neuroscience; neural; mechanism
MeSH Terms: conditions — Parkinson Disease; Movement Disorders

ARMS (1):
- PK-16CH EXG system (Experimental): PK-16CH EXG is a wireless physiological signal acquisition system for monitoring the bio-signals, such as EEG, ECG, and EMG. The system can concomitant EEG and EMG recording during ambulation.
  Interventions: Device: PK-16CH EXG system

INTERVENTIONS:
Device: PK-16CH EXG system

SUMMARY:
We aim to investigate the higher level mechanism of gait disorders in PD patients by ambulatory recording of electroencephalographic (EEG) and leg electromyographic (EMG) signals during unconstrained walking. Independent component analysis will be conducted for signal analysis. The connectivity among different brain regions will also be investigated. The PD patients received deep brain stimulation will be recruited for the study. The local field potentials recorded from sub-thalamic nuclei and/or PPN will be recorded concomitantly with EEG and leg EMG signals during unconstrained walking in PD patients to assess the roles of these deep structures in ambulation and their functional connectivity with other brain regions during walking.

DETAILED DESCRIPTION:
Gait disorder in Parkinson's disease (PD) contains several aspects including particularly the slowness of walking and freezing of gait (FOG). These problems may sometimes cause fall of patients and culminate in severe head injury and bony fracture. In this regard the understanding of freezing of gait and other parkinsonian ambulatory disorders is important for the management of patients. Previous electrophysiological studies of gait disorders were majorly focused on the kinetic and kinematric measurements. How the higher level neural structures including the cerebral cortex, basal ganglia, sub-thalamic nucleus or pedunculopontine nucleus were involved in the gait processing are currently unknown. A recent study by adopting movement related cortical potential (MRCP) recording to probe the PD ambulatory disorders in freezing and non-freezing patients illustrated that PD patients with FOG lost the relationship between stride length and the movement related potentials. Since the study was performed in constrained condition and each trigger for MRCP did not guarantee to be of freezing nature in FOG patients, the results cannot reflect the true manifestations of gait freezing in PD patients. In the current proposal, we will perform concomitant recording of the scalp electroencephagraphic and leg electromyographic signals during unconstrained walking in normal subjects and PD with or without FOG. Independent component analysis (ICA) will be conducted for analyzing the possible differences of patterns among the three groups and within the FOG patients during the freezing and non-freezing phases. In addition, the cortical effective connectivity among different cortical regions during freezing and non-freezing phase will also be assessed. Since sub-thalamic nuclei and pedunculopontine nucleus may be involved in the ambulatory circuitry, we will also investigate this possibility in PD patients to be treated with deep brain stimulation. The nuclear local field potentials will be recorded concomitantly with scalp electroencephalographic signals and electromyographic signals during unconstrained signals. ICA and event related de-synchronization analysis will be conducted to understand the roles of these nuclei in walking. The effective connectivity of the deep nuclei and the cortical regions will also be assessed to learn the functional set of ambulation. The pioneer exploration of the higher level neural manifestations of walking will extend the spectrum from conventional kinetic and kinematric gait analysis to peep how the central neural circuitry operate in ambulation.

ELIGIBILITY:
Inclusion Criteria:

Patients with PD will be diagnosed according to the Brain Bank criteria.

Exclusion Criteria:

1. impairment of cognition that leads unable to fully cooperate with the oral commands during operation.
2. any moderate to severe medical disorders such as poor control of diabetic mellitus, functional III or above congestive heart failure, or cancer with distant metastasis etc.
3. severe mood disorders such as major depression.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2014-08; Primary Completion 2015-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Recording of electroencephalographic (EEG) and electromyographic (EMG) signals during unconstrained walking. | Baseline
  Variables in gait analysis:1.Gait initiation; 2.Level walking; 3.Turning; 4.Gait termination.

SECONDARY OUTCOMES:
Unified Parkinson's Disease Rating Scale (UPDRS) | Baseline
  The UPDRS score has three parts, part I (Mentation, Behavior and Mood), Part II (Activities of Daily Living) and Part III (Motor Examination). Each consisting of questions answered on a 0-4 point scale. The minimum total score possible is 0 and the maximum total score possible is 176. Higher scores indicating more severe symptoms.
The 39-item Parkinson's Disease Questionnaire (PDQ-39) | Baseline
  The PDQ-39 contains 39-items covering 8 discrete dimensions: mobility, activities of daily living, emotional well-being, stigma, social support, cognitions, communication, and bodily discomfort. Each question is scored on a 5-point scale and recoded to 0 to 4 for the analysis. The total score can range from 0 to 132 and with a higher score indicating more severe symptoms.
The Fall Assessment Test of CMUH | Baseline
Tinetti Performance Oriented Mobility Assessment (POMA) | Baseline
  The Tinetti assessment tool is an easily administered task-oriented test that measures an older adult's gait and balance abilities. The total score can range from 0 to 28 and with a lower score indicating more severe symptoms.
New freezing of gait questionnaire (NFOG-Q) | Baseline
  The New Freezing of Gait Questionnaire (NFOG-Q) is a clinician-administered tool that aims to assess both the clinical aspects of FOG as well as its subsequent impairments on quality of life.
Mini-Mental State Examination (MMSE) | Baseline
  MMSE consists of five sections (orientation, registration, attention-calculation, recall, and language) and results in a total possible score of 30, with higher scores indicating better function.

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital/Neuro Depart, Taichung, Taiwan, Taiwan